CLINICAL TRIAL: NCT05054114
Title: Prospective Randomized Open-label Comparative Study of the Use of Intranasal Form of Interferon Gamma Human Recombinant in Patients for the Prevention of Acute Respiratory Viral Infections, Including COVID-19
Brief Title: Study of the Use of Nasal IFN-γ in Patients for the Prevention of Acute Respiratory Viral Infections, Icluding COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPP Pharmaclon Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RAIN-2020
Record Dates: First submitted 2021-09-21; First posted 2021-09-23 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2021-09

CONDITIONS: COVID-19 Respiratory Infection; Acute Respiratory Disease
Keywords: COVID-19 prevention, interferon gamma, nasal drops

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug: Interferon Gamma (Experimental): IFN-G administered for 2 10-day courses with a 1-week pause between the courses.
  Interventions: Drug: Interferon gamma human recombinant (IFN-G)
- Control: No intervention (No Intervention): Any preventive method including a variety of pharmacologic therapies against COVID-19, alongside the use of antiviral and immunomodulating agents, with the exception of drugs prescribed off-label or for research purposes, and IFN-G as well.

INTERVENTIONS:
Drug: Interferon gamma human recombinant (IFN-G) — nasal form
  Other Names: Ingaron
  Arms: Drug: Interferon Gamma

SUMMARY:
It is known that the pretreatment with exogenous interferon blocks SARS-CoV-2 infection, but intervention is much more effective if administered prior to infection. In this study the primary aim is to investigate 28-day regime of nasal interferon gama use in healthy participants for COVID-19 and other respiratory infections prevention.

DETAILED DESCRIPTION:
The tissues of the upper respiratory tract: the mucous membrane of the oropharynx, nose, - as well as the lung parenchyma are identified as the main targets of SARS-CoV-2. Previously published data from studies describe that in vitro and in vivo observations SARS-CoV-2 replicates exponentially during the first few days after infection to the peak of the host's antiviral response. It is assumed that it is the violation of the antiviral immunity of the nasal epithelium that may underlie the development of a severe form of the disease. The significance of interferon protection proven in early studies supposes that it can reduce peak viral load and viral reproduction index.

To confirm the efficacy and safety of nasal interferon gama use in healthy participants for COVID-19 and other respiratory infections prevention there is a need of interventional study. Interferon gamma has many years of clinical experience in the prevention and treatment of various viral infections, including coronavirus nature, flu and pneumonia.

After participant enrollment, comprehensive baseline documentation of anamnestic, clinical and allergy data is collected on the same day if possible. For participants who develops acute respiratory symptoms or recieve positive PCR test for SARS-CoV-2, all parameters are collected that may be necessary to assess the type and severity of acute respiratory disease. Furthermore, data is collected that may be suitable for an assessment of the safety profile. In particular, questions are asked about known infection risks, lifestyle, alternative prevention methods, immune competence, rate of acute respiratory infections, the history of symptoms and tests relating to COVID-19, preexisting medication, as well as ethnicity.

On the day of inclusion (day -3-1) routine clinical values, safety-relevant data, WHO scale score, concomitant medication and anamnesis, as well as study criteria analysis are documented.

On the day 0 (randomization visit) and at termination visit (up to 90 days) repeated routine clinical values, safety-relevant data, WHO scale score, and concomitant medication are collected. If the patient falls ill, the necessary disease information is documented. If the patient dies, the date and cause of death are documented.

On days 24-30 after randomization, a follow-up call takes place with particular attention to the health-related events such as respiratory diseases or other changes in health and vital status and drug compliance. If the participant cannot be reached for the follow-up call, the including study center will attempt to reach the participant, otherwise exclude the participant.

A nasopharynx swab is obtained on days 0 to exclude asymptomatic patients before the randomisation. If possible, sputum is obtained for termination visit and during the acute respiratory symproms manifestation to confirm COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of both sexes over 18 years of age.
* Obtaining written informed consent.
* Ability and consent to participate in this research.
* Absence of symptoms of respiratory infection.
* A negative result of a PCR study for the presence of RNA SARS-CoV-2 according to biomaterial obtained by nasopharyngeal smear.

Exclusion Criteria:

* Any other concomitant diseases or conditions, which, in the opinion of the research doctor, may distort research results, restrict the rights of a volunteer or put him/her at greater risk.
* Contraindications to the use of the investigated medicinal product.
* Individual intolerance to the ingredients included in the composition of the investigational medicinal product.
* Pregnancy or breastfeeding.
* Doubtful result of a PCR test for the presence of RNA SARS-CoV-2 in the biomaterial obtained by nasopharyngeal smear.
* Participation in a clinical trial using study therapy within 30 days prior to enrollment in this study.
* Disagreement to follow in the research reliable contraceptive measures (abstinence; or a combination of 2 different methods: for example, barrier and spermicides, or barrier and intrauterine device, or barrier and hormonal, etc.) - for participants with saved reproductive potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly I Saulin, Master, Study Director — SPP Pharmaclon Ltd.
Locations (1):
- City Clinical Hospital named after M.E. Zhadkevich Moscow City Health Department, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug: Interferon Gamma | Control: No Intervention
Started | 315 | 315
Completed | 302 | 313
Not Completed | 13 | 2
Not completed — Protocol Violation | 13 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug: Interferon Gamma | Control: No Intervention | Total
Number analyzed (Participants) | 315 | 315 | 630
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 305 | 299 | 604
  >=65 years | 10 | 16 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 117 | 232
  Male | 200 | 198 | 398
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 56 | 61 | 117
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 259 | 254 | 513
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 315 | 315 | 630
Vaccination against COVID-19 [Number; unit: Participant] | 57 | 74 | 131

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients With Acute Respiratory Viral Infections, Including COVID-19, at the End of the Prophylactic Period
Description: The proportion of patients with acute respiratory viral infections, including COVID-19, assessed at visit 2 (at the end of the prophylaxis course and before the start of the follow-up period)
Time Frame: 28 days
Population: The results of the assessment of the incidence rate at the end of the prophylaxis period
Measure: Number; unit: participants
Arm/Group | Drug: Interferon Gamma | Control: No Intervention
Number analyzed (Participants) | 315 | 315
participants | 3 | 13

2. Secondary Outcome: The Proportion of Patients With Confirmed COVID-19 at the End of the Prophylactic Period
Description: The proportion of patients with COVID-19, assessed at visit 2 (at the end of the prophylaxis course and before the start of the follow-up period)
Time Frame: 28 days
Population: The results of the assessment of the incidence of COVID-19 at the end of the prevention period
Measure: Number; unit: participants
Arm/Group | Drug: Interferon Gamma | Control: No Intervention
Number analyzed (Participants) | 315 | 315
participants | 0 | 0

3. Secondary Outcome: The Proportion of Patients With Acute Respiratory Viral Infections, Including COVID-19, at the End of the Follow-up Period
Description: The proportion of patients with acute respiratory viral infections, including COVID-19, assessed at visit 3 (at the end of the study)
Time Frame: 2 months
Population: The results of the assessment of the incidence rate at the end of the study
Measure: Number; unit: participants
Arm/Group | Drug: Interferon Gamma | Control: No Intervention
Number analyzed (Participants) | 315 | 315
participants | 6 | 25

4. Secondary Outcome: Proportion of Patients With Confirmed COVID-19 at the End of the Follow-up Period
Description: The proportion of patients with COVID-19, assessed at visit 3 (at the end of the study)
Time Frame: 2 months
Population: The results of the assessment of the incidence of COVID-19 at the end of the prevention period
Measure: Number; unit: participants
Arm/Group | Drug: Interferon Gamma | Control: No Intervention
Number analyzed (Participants) | 315 | 315
participants | 0 | 2

5. Secondary Outcome: Number of Participants With a Complicated Course of Infection
Description: The rate of complicated courses of infection among cases
Time Frame: 2 months
Population: The results of assessing the frequency of complicated course
Measure: Number; unit: participants
Arm/Group | Drug: Interferon Gamma | Control: No Intervention
Number analyzed (Participants) | 315 | 315
participants | 0 | 0

6. Secondary Outcome: The Proportion of Participants With Each Score of the WHO Clinical Improvement Scale
Description: The proportion of participants with each score (0-8) on the WHO Clinical Improvement Scale from 0 points - not infected, no manifestations or virological signs of infection, up to 8 points - died, death
Time Frame: 28 days
Population: The results of assessing the frequency of different scores on the WHO scale at the end of the prophylaxis period
Measure: Number; unit: participants
Arm/Group | Drug: Interferon Gamma | Control: No Intervention
Number analyzed (Participants) | 3 | 13
participants
  0 points on the WHO scale | 0 | 0
  1 points on the WHO scale | 3 | 13
  2 points on the WHO scale | 0 | 0
  3 points on the WHO scale | 0 | 0
  4 points on the WHO scale | 0 | 0
  5 points on the WHO scale | 0 | 0
  6 points on the WHO scale | 0 | 0
  7 points on the WHO scale | 0 | 0
  8 points on the WHO scale | 0 | 0

7. Secondary Outcome: The Proportion of Participants With Each Score of the WHO Clinical Improvement Scale
Description: as for outcome 6
Time Frame: 2 months
Population: The results of assessing the frequency of different scores on the WHO scale at the end of the prophylaxis period
Measure: Number; unit: participants
Arm/Group | Drug: Interferon Gamma | Control: No Intervention
Number analyzed (Participants) | 6 | 26
participants
  0 points on the WHO scale | 0 | 0
  1 points on the WHO scale | 6 | 25
  2 points on the WHO scale | 0 | 1
  3 points on the WHO scale | 0 | 0
  4 points on the WHO scale | 0 | 0
  5 points on the WHO scale | 0 | 0
  6 points on the WHO scale | 0 | 0
  7 points on the WHO scale | 0 | 0
  8 points on the WHO scale | 0 | 0

8. Secondary Outcome: The Duration of Symptoms in Participants With Acute Respiratory Viral Infections, Including COVID-19
Description: The duration of symptoms in participants with acute respiratory viral infections, including COVID-19, assessed at the end of the study
Time Frame: 2 months
Population: Duration of disease symptoms at the end of the study (2 months)
Measure: Median (Full Range); unit: days
Arm/Group | Drug: Interferon Gamma | Control: No Intervention
Number analyzed (Participants) | 3 | 13
days | 4.17 [2.00 to 8.00] | 6.76 [1.00 to 24.00]

9. Secondary Outcome: The Duration of Symptoms in Participants With Acute Respiratory Viral Infections, Including COVID-19
Description: The duration of symptoms in participants with acute respiratory viral infections, including COVID-19, assessed at the end of prevention course
Time Frame: 28 days
Population: Duration of disease symptoms at the end of the prophylaxis period (28 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Drug: Interferon Gamma | Control: No Intervention
Number analyzed (Participants) | 3 | 13
days | 5.33 [2.00 to 8.00] | 4.15 [1.00 to 8.00]

ADVERSE EVENTS:
Time Frame: Safety assessment was carried out throughout the observation period, starting from the inclusion of the participant in the study - within 2 months.
Description: No serious adverse events or reactions were reported during the study.
Arm/Group | Drug: Interferon Gamma | Control: No Intervention
All-Cause Mortality (participants affected / at risk) | 0/315 | 0/315
Serious Adverse Events (participants affected / at risk) | 0/315 | 0/315
Other Adverse Events (participants affected / at risk) | 24/315 | 21/315
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug: Interferon Gamma (N=315) | Control: No Intervention (N=315)
Headache (Nervous system disorders) | 11 (11) | 8 (8)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Increase in blood pressure (Vascular disorders) | 4 (4) | 3 (3)
Joint pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin hardening (Infections and infestations) | 1 (1) | 0 (0)
Lower abdominal pain (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rashes on the nasal mucosa (herpetic) (Infections and infestations) | 0 (0) | 2 (2)
Frequent urination (Renal and urinary disorders) | 0 (0) | 1 (1)
Increasing PSA levels (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pain when urinating (exacerbation of chronic prostatitis) (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT05054114/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT05054114/SAP_001.pdf